CLINICAL TRIAL: NCT07386782
Title: Palpatory and Ultrasonographic Assessment of Tissue Compressibility: Validation and Learning Effects in Phantom Models
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: Req-2025-01655
Record Dates: First submitted 2026-01-20; First posted 2026-02-04 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Exanimation; Diagnostic Ultrasound; Palpation
Keywords: Exanimation; Diagnostic Ultrasound; Palpation
MeSH Terms: conditions — Coma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: Ultrasonographic Compression Measurment and Palpation of Standardized Phantom Models — Repeated ultrasonographic compression measurements and palpation of standardized phantom models

SUMMARY:
This validation study compares clinical palpation and ultrasonographic measurements of tissue compressibility using standardized phantom models. Operators with different levels of clinical and ultrasound experience perform repeated, blinded assessments across multiple sessions. The study evaluates accuracy, reliability, agreement between modalities, and learning effects over time, aiming to support standardized and more objective assessment of tissue compressibility in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Medical professionals and medical students

Exclusion Criteria:

* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with different years of clinical experience and levels of experience in ultrasound diagnostics (medical students, residents, and attendings) will be included. Age >= 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy and reliability of palpation and ultrasonographic compression measurements | Over 3 sessions, seperated by at least 1 day and at most 1 week (study duration: 3 days to 2 weeks)
  Intraoperator and interoperator accuracy and reliability of palpation and ultrasonographic compression measurements on two phantom models as intraclass correlation coefficient and linear mixed-effects model

SECONDARY OUTCOMES:
Effect of operator characteristics on the measurement accuracy and reliability. | Over 3 sessions, seperated by at least 1 day and at most 1 week (study duration: 3 days to 2 weeks)
  Operator characteristics (age, gender, level of experience) will be introduced as fixed effects in a linear mixed-effects model with a random effect for participants to account for repeated measurements
Assess the learning curve in palpation and ultrasound measurements | Over 3 sessions, seperated by at least 1 day and at most 1 week (study duration: 3 days to 2 weeks)
  Changes in accuracy of both modalities using linear mixed-effects model with a random effect for participants to account for repeated measurements. To test possible confounding factors, they will be introduced as fixed effects.
Correlate the compression measurements with palpatory assessment | Over 3 sessions, seperated by at least 1 day and at most 1 week (study duration: 3 days to 2 weeks)
  Correlation of both modalities using linear mixed-effects model with a random effect for participants to account for repeated measurements. To test possible confounding factors, they will be introduced as fixed effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Inselspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The data supporting this study's findings are available upon request from Samuel Tschopp, the corresponding author.
Supporting Information: Study Protocol, SAP, Analytic Code
Access Criteria: The data supporting this study's findings are available upon request from Samuel Tschopp, the corresponding author.